CLINICAL TRIAL: NCT06524011
Title: Split Face Comparative Study of Stromal Vascular Fraction Enriched PRP Versus Each Alone in Treatment of Atrophic Post-acne Scars
Brief Title: Stromal Vascular Fraction Enriched PRP in Treatment of Post-acne Scars
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mona El Radi Kamal Mohamed Emam, Dermatology assistant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dr. MonaRadi
Record Dates: First submitted 2023-10-06; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Acne Scars - Atrophic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SVF enriched PRP vs PRP (Experimental)
  Interventions: Biological: Stromal vascular fraction (SVF) enriched platelet rich plasma (PRP) versus each alone
- SVF enriched PRP vs SVF (Active Comparator)
  Interventions: Biological: Stromal vascular fraction (SVF) enriched platelet rich plasma (PRP) versus each alone
- PRP vs SVF (Active Comparator)
  Interventions: Biological: Stromal vascular fraction (SVF) enriched platelet rich plasma (PRP) versus each alone

INTERVENTIONS:
Biological: Stromal vascular fraction (SVF) enriched platelet rich plasma (PRP) versus each alone — Adipose derived stromal vascular fraction cells will be aspirated and isolated from patient autologous adipose tissue and used to enrich patient's autologous platelet rich plasma then will be used to treat atrophic post acne scars versus each alone.

SUMMARY:
in a split face fashion, 30 patients will be randomized into 3 groups: Group A: rt side treated with SVF enriched PRP, lt side treated with prp Group B: rt side treated with SVF enriched PRP, lt side treated with SVF Group C: rt side treated with PRP, lt side treated with SVF

ELIGIBILITY:
Inclusion Criteria:

* patients with atrophic post acne scars without any previous treatment trials.
* adequate blood picture, no anemia, no bleeding or platelet disorders.

Exclusion Criteria:

* pregnant and lactating females.
* elderly.
* patients with bleeding tendencies.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
change in severity of acne scars using Goodman scoring system | 3 monthly sessions and follow up for 3 months after the last visit
  at baseline, acne scars will be assessed clinically using the 4 point grading system proposed by Goodman &colleagues in 2006, patients' complaints and expectations will be addressed as well and the impact of acne scars on patients' quality of life will be investigated using the dermatology life quality index (DLQI). Goodman scoring system will be used at the last session and at the follow up visit to measure the change pre and post treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Hospitals, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: Undecided